CLINICAL TRIAL: NCT00231764
Title: Evaluating Safety and Efficacy of MMF, Daclizumab and Corticosteroids as Mainstay Immunosuppression in Combination With Low-Dose CsA, Tac or Sir in Comparison to Current Standard Immunosuppression (MMF, CsA and Corticosteroids) in Renal Tx
Brief Title: MMF, Daclizumab and Corticosteroids as Mainstay Immunosuppression in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ekberg, Henrik, M.D. (Individual)
Collaborators: Prof. Philip Halloran, Edmonton, Canada (sponsor) (Unknown); Prof. Yves Vanrenterghem, Leuven, Belgium (Steering Committee Member) (Unknown); Prof. Pierre Daloze, Montréal, Canada (Steering Committee Member) (Unknown); Prof. Thomas C. Pearson, Atlanta, USA (Steering Committee Member) (Unknown); Prof. Ulrich Frei, Berlin, Germany (Steering Committee Member) (Unknown); Prof. Flavio Vincenti, San Francisco, USA (Ass. Steering Committee Member) (Unknown); Prof. Josep Grinyo, Barcelona, Spain (Ass. Steering Committee Member) (Unknown); Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SYMPHONY
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Kidney Transplantation
Keywords: Renal transplantation; Immunosuppression; Daclizumab; GFR
MeSH Terms: interventions — Daclizumab

INTERVENTIONS:
Drug: daclizumab

SUMMARY:
To determine the renal function, as expressed by the glomerular filtration rate at 12 months, in renal transplant recipients receiving mycophenolate mofetil, daclizumab, and corticosteroids as mainstay immunosuppression in combination with low-dose cyclosporine, tacrolimus, or sirolimus, and compare it to that of renal transplant recipients receiving standard immunosuppression with mycophenolate mofetil, normal dose cyclosporine and corticosteroids.

DETAILED DESCRIPTION:
The purpose of the SYMPHONY study is to compare four different immunosuppressive regimens. They are each given for one year. The following four combinations are tested in four groups of patients:

* Group A: Cyclosporine in a normal dosage, mycophenolate mofetil (MMF) and corticosteroids
* Group B: Daclizumab in the first two months after transplantation, cyclosporine in a lower dosage compared to group A, mycophenolate mofetil (MMF) and corticosteroids
* Group C: Daclizumab in the first two months after transplantation, tacrolimus in low dosage, mycophenolate mofetil (MMF) and corticosteroids
* Group D: Daclizumab in the first two months after transplantation, sirolimus in a low dosage, mycophenolate mofetil (MMF) and corticosteroids.

All drugs of the four immunosuppressive regimes are approved by the Health Authorities in the participating country for use in kidney transplantation. The regimen administered to the patients in Group A represents a standard treatment, currently given with success to many transplant patients in a number of countries in the world. The treatments in Groups B, C and D are experimental in the sense that either the doses administered are lower than the ones used before and/or the combination of drugs is experimental. Nevertheless, there are results of scientific studies indicating that they are all effective alternatives and that they might have advantages compared to the standard immunosuppressive regimen, in particular as far as their safety (side effects, long-term toxicity) is concerned. However, from the previous clinical experience, it is not yet clear which regimen offers the most advantages for the patients. To find this out, in SYMPHONY the four regimens are administered to the four groups of patients (A-D) and the results in the different groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 - 75 years
* Recipients of single-organ renal primary allograft or second renal transplants (provided that the previous graft was not lost from acute rejection within the first year) from living or cadaver donors
* Patients who provide written informed consent.

Exclusion Criteria:

* PRA > 20% within 6 months prior to enrollment
* Cold ischemia time > 30 hours
* Previous treatment with daclizumab
* History of malignancy (except localized skin cancer)
* Active peptic ulcer disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1760
Dates: Start 2002-11; Primary Completion 2006-05 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
GFR calculated from the serum creatinine with the Cockcroft-Gault formula at 12 months posttransplantation

SECONDARY OUTCOMES:
Acute rejection rate at 6 and 12 months, patient and graft survival rates at 12 months
Treatment failure during the first twelve months
Time to first acute rejection
Patient and graft survival at 6 and 12 months posttransplant
Calculated GFR using the Cockcroft-Gault formula during the study and measured GFR at month 12
Incidence of Delayed Graft Function (DGF)
Safety Parameters:
Clinical assessments, vital signs, laboratory analyses, adverse events, opportunistic infections, malignancies, and deaths
Incidence of failure to achieve primary closure of transplant surgical wound at 2 weeks
Incidence of lymphocele requiring intervention in the first 6 months posttransplant

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Ekberg, Prof., Study Chair — Malmo University Hospital, Malmö, Sweden; Philip Halloran, Prof., Study Chair — University of Alberta, Edmonton, Canada

REFERENCES:
- [Derived] Ekberg H, Tedesco-Silva H, Demirbas A, Vitko S, Nashan B, Gurkan A, Margreiter R, Hugo C, Grinyo JM, Frei U, Vanrenterghem Y, Daloze P, Halloran PF; ELITE-Symphony Study. Reduced exposure to calcineurin inhibitors in renal transplantation. N Engl J Med. 2007 Dec 20;357(25):2562-75. doi: 10.1056/NEJMoa067411. PMID 18094377